CLINICAL TRIAL: NCT01220882
Title: Skeletal Age Assessment From the Olecranon For Slipped Capital Femoral Epiphysis
Brief Title: Evaluation of Skeletal Maturity for Slipped Capital Femoral Epiphysis
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Rutgers, The State University of New Jersey (Other)
Responsible Party: Principal Investigator, bone123, Assistant Professor, Rutgers, The State University of New Jersey
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 0120080287
Record Dates: First submitted 2010-08-19; First posted 2010-10-14 (Estimated); Last update posted 2013-12-25 (Estimated); Status verified 2013-12

CONDITIONS: Slipped Capital Femoral Epiphysis
Keywords: Slipped capital femoral epiphysis
MeSH Terms: conditions — Slipped Capital Femoral Epiphyses

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Radiographic skeletal age assessment (No Intervention): Participant group studied will include all pediatric patients presenting to our institution with a unilateral or bilateral SCFE. Patients with metabolic and endocrine conditions will be included.
  Interventions: Radiation: Radiographic skeletal age assessment

INTERVENTIONS:
Radiation: Radiographic skeletal age assessment — bone age assessment from the elbow lateral radiograph

SUMMARY:
This study is being done for two reasons: 1) to evaluate growth problems in the hip in patients with Slipped Capital Femoral Epiphysis (SCFE) as they continue to grow into adults, and 2) to help doctors determine which patients are at risk for developing a SCFE on their opposite hip. Studies show that up to 60% of patients with a SCFE will go on to develop a SCFE on their other side. Being able to better determine which patients are at risk for developing a SCFE on the other side will help physicians better monitor patients with a history of a SCFE and perhaps treat them before they develop a SCFE on the opposite side. By studying the growth centers seen on X-rays of your child's legs and elbow, the investigators may be able to better predict which children with a SCFE are at risk for developing a SCFE on their opposite hip and potential growth problems as they continue to grow.

DETAILED DESCRIPTION:
After obtaining informed consent, pediatric patients presenting to our institution with a SCFE will have a single radiograph of the elbow, in addition to those radiographs currently obtained as part of routine evaluation and treatment (e.g. AP pelvis, bilateral hip laterals, scanogram, and hand bone age). This additional radiograph, a single one-time lateral elbow radiograph taken on initial presentation with a SCFE, will be used to assess bone age and compared with other radiographic methods, i.e. hand bone age, currently used to assess skeletal maturity. Scanogram of the lower extremities, at initial presentation and at the completion of skeletal growth, will be used to accurately assess the length of the lower extremities and evaluate limb length discrepancy at maturity. Treatment of the patient's SCFE and post-operative management will be as per routine care at our institution. Patients will be followed until skeletal maturity.

The medical records and radiographs of patients with SCFE will be collected. Patient data will include:

* Patient demographics- chronologic age, gender, race/ethnicity, standing height, weight, BMI, clinical follow-up duration
* SCFE type- chronicity of symptoms prior to presentation, Loder classification of slip stability, laterality, time between sequential SCFEs
* Skeletal maturity data- bone age, triradiate closure, Risser sign, modified Oxford bone age, olecanon method and the Simplified skeletal maturity scoring system
* Radiographic data- slip severity, physeal slope angle, and leg length discrepancy
* Complications
* Additional procedures

In order to compare the various radiographic methods of skeletal age assessment, the elbow hand and AP pelvis radiographs will be reviewed once by three independent and experienced observers, two pediatric orthopaedic surgeons and one musculoskeletal radiology attending. The radiographic skeletal age assessment will be discussed by these three observers in order to minimize intraobserver and interobserver errors.

ELIGIBILITY:
Inclusion Criteria:

* Slipped capital femoral epiphysis

Exclusion Criteria:

* Prior Slipped capital femoral epiphysis not initially treated at our institution

Ages: 8 Years to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 60 (Estimated)
Dates: Start 2008-10; Primary Completion 2015-07 (Estimated); Study Completion 2015-12 (Estimated)

PRIMARY OUTCOMES:
Radiographic data on skeletal maturity and SCFE radiographic characteristics | Day 1
  Radiographic assessment on initial presentation of SCFE on hip and pelvis x-rays, limb length discrepancy on Scanogram, and bone age measurement using hand AP radiograph and lateral view of the elbow.

SECONDARY OUTCOMES:
Clinical examination | Year 8
  Skeletal maturity will be determined when the proximal femoral physis have both fused (approximately age 14 years for girls and 16 years for boys).
Radiographic evaluation of Limb length discrepancy on Scanogram | Year 8
  Skeletal maturity will be determined when the proximal femoral physis have both fused (approximately age 14 years for girls and 16 years for boys).

CONTACTS AND LOCATIONS:
Overall Officials: Tamir Bloom, MD, Principal Investigator — Rutgers University
Locations (1):
- University of Medicine and Dentistry of New Jersey, Newark, New Jersey, United States